CLINICAL TRIAL: NCT04940871
Title: A Randomized, Double-blind, Placebo-controlled Study to Assess the Efficacy and Safety of Favipiravir-HU Compared to Placebo as add-on Therapy to Standard of Care in Asymptomatic to Mild Severity COVID-19 Patients
Brief Title: Study to Assess the Efficacy and Safety of Favipiravir-HU
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Only one patient was enrolled, who who later withdrew the consent. They decided not to contunie the study.
Sponsor: University of Pecs (Other)
Collaborators: Hungarian Ministry of Innovation and Technology (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HUN-FAVI-02
Record Dates: First submitted 2021-05-20; First posted 2021-06-28 (Actual); Last update posted 2022-11-09 (Actual); Status verified 2022-11

CONDITIONS: Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2)
MeSH Terms: interventions — Hardness

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: double-blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Favipiravir HU + SOC (Experimental): Favipiravir HU + SOC
  Interventions: Drug: Favipiravir HU 200 mg hard capsules
- Placebo HU + SOC (Placebo Comparator): Placebo HU + SOC
  Interventions: Drug: Placebo HU

INTERVENTIONS:
Drug: Favipiravir HU 200 mg hard capsules — Drug substance: Favipiravir Dose: 200 mg Administration: oral Formulation: capsules
  Arms: Favipiravir HU + SOC
Drug: Placebo HU — Name: Placebo clinical sample Drug substance: placebo Dose: - Administration: oral Formulation: capsules
  Arms: Placebo HU + SOC

SUMMARY:
The aim of the study is to assess the safety and efficacy of Favipiravir HU when administered to SARS-Cov- 2 patients in order to offer a safe and effective treatment to SARS-Cov-2 infection during the pandemic. The study is not for registration purposes and is not part of a series of studies for registration of Favipiravir HU.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients between the ages of 18 and 65 years.
2. Patients with PCR confirmed SARS-CoV-2 infection
3. Asymptomatic or have mild only symptoms and symptoms are onset less than 5 days
4. Signed Informed Consent Form and Patient Information Leaflet

Exclusion Criteria:

1. Pregnant or possibly pregnant patients or lactating females
2. Patients have moderate to severe or immediately life-threatening COVID-19
3. Major risk factor onset (Obesity, Diabetes, COPD, Hypertension)
4. Patients with SpO2 less than 95% without oxygen therapy
5. Patients with severe hepatic impairment equivalent to Grade C on Child-Pugh classification
6. Patients with renal impairment requiring dialysis
7. Patients with disturbed consciousness such as disturbed orientation
8. Female patients who are woman of childbearing potential and unable to consent to use of dual contraception from the start of favipiravir administration to 30 days after the end of favipiravir administration. Dual contraception is a combination of two of the following: Barrier method of contraception: condoms (male or female) with orwithout a spermicidal agent, diaphragm or cervical cap with spermicide; IUD; Hormone-based contraceptive; Tubal ligation
9. Male patients whose are unable to consent to use of barrier method of contraception (condom) the start of favipiravir administration to 90 days after the end of favipiravir administration. Male patients who are planning to donate sperm in 90 days after the start of favipiravir administration.
10. Patients with hereditary xanthinuria
11. Patient with severe uncontrolled hyperuricaemia
12. Patients receiving immunosuppressants
13. Patients who received interferon-alpha or drugs with reported antiviral activity against SARS-CoV- 2 (hydroxychloroquine sulfate, chloroquine phosphate, lopinavir-ritonavir combination, ciclesonide, nafamostat mesylate, camostat mesylate, remdesivir, etc.) within 72 hours or Patients who receive forbidden concomitant medication
14. Any medical condition that the examining physician deems unsuitable for the patient to participate in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2021-11-25 (Actual); Primary Completion 2021-11-29 (Actual); Study Completion 2021-11-29 (Actual)

PRIMARY OUTCOMES:
PRIM1_ the percentage of virus copy number | 5 months
  The primary endpoint of the study is the percentage of virus copy number at Day6 compared to baseline.

SECONDARY OUTCOMES:
SEC1_mortality rate | 6 months
  Overall mortality rate
SEC2_respiratory failure | 6 months
  Proportion of patients with respiratory failure
SEC3_ intensive care | 6 months
  Proportion of patients with need for intensive care
SEC4_non-invasive respiratory support | 6 months
  Proportion of patients with need for non-invasive respiratory support
SEC5_ invasive respiratory support | 6 months
  Proportion of patients with need for invasive respiratory support
SEC6_ Acute Respiratory Distress Syndrome | 6 months
  Proportion of patients with Acute Respiratory Distress Syndrome

OTHER OUTCOMES:
KSEC1_Time to virus elimination | 5 months
  Number of days from treatment start to virus elimination
KSEC2_severe stages of COVID-19 | 6 months
  Proportion of patients achieving more severe stages of COVID-19
KSEC3_Time to recovery | 6 months
  Time to recovery in patients who have developed symptoms
KSEC4_ adverse event | 6 months
  Number and proportion of patients with at least 1 adverse event related to study treatment

CONTACTS AND LOCATIONS:
Locations (1):
- University of Szeged - Internal Medicine, Szeged, Hungary

IPD SHARING:
Plan to Share IPD: Undecided